CLINICAL TRIAL: NCT01994993
Title: Antibiotic Safety in Infants With Complicated Intra-Abdominal Infections (SCAMP Trial)
Brief Title: Antibiotic Safety (SCAMP)
Acronym: SCAMP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Michael Cohen-Wolkowiez (Other)
Collaborators: The Emmes Company, LLC (Industry)
Responsible Party: Sponsor-Investigator, Michael Cohen-Wolkowiez, Associate Professor, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00048773; HHSN275201000003I (Other Grant/Funding Number: NICHD)
Record Dates: First submitted 2013-11-18; First posted 2013-11-26 (Estimated); Results first posted 2018-02-27 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Complicated Intra Abdominal Infections
Keywords: Antibiotics; ampicillin; metronidazole; clindamycin; piperacillin-tazobactam; Safety; Infants; Intra abdominal infections
MeSH Terms: conditions — Intraabdominal Infections | interventions — Ampicillin; Metronidazole; Gentamicins; Clindamycin; Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group 1 (ampicillin +gentamycin +metronidazole) (Active Comparator): Ampicillin and gentamycin and metronidazole
  Interventions: Drug: ampicillin and metronidazole and gentamicin
- Group 2 (ampicillin +gentamicin+clindamycin) (Active Comparator): ampicillin and gentamicin and clindamycin
  Interventions: Drug: ampicillin and gentamicin and clindamycin
- Group 3 (piperacillin-tazobactam and gentamicin) (Active Comparator): piperacillin-tazobactam and gentamicin
  Interventions: Drug: gentamicin and Piperacillin- tazobactam
- Group 4 (metronidazole) (Active Comparator): Per standard of care antibiotics, and Metronidazole
  Interventions: Drug: standard of care antibiotics and metronidazole
- Group 5 (metronidazole/clindamycin/piperacillin-tazobactam) (Active Comparator): metronidazole, clindamycin, or piperacillin-tazobactam
  Interventions: Drug: metronidazole, clindamycin, or piperacillin-tazobactam

INTERVENTIONS:
Drug: ampicillin and metronidazole and gentamicin — IV infusion of ampicillin and metronidazole and gentamicin for a total of 10 days. Dose based on postnatal age (PNA) and gestational age(GA)
  Arms: Group 1 (ampicillin +gentamycin +metronidazole)
Drug: ampicillin and gentamicin and clindamycin — IV infusion of ampicillin and gentamicin and clindamycin for a total of 10 days. Dose based on postnatal age (PNA) and gestational age(GA)
  Arms: Group 2 (ampicillin +gentamicin+clindamycin)
Drug: gentamicin and Piperacillin- tazobactam — IV infusion of gentamicin and Piperacillin- tazobactam for a total of 10 days. Dose based on postnatal age (PNA) and gestational age(GA)
  Arms: Group 3 (piperacillin-tazobactam and gentamicin)
Drug: standard of care antibiotics and metronidazole — IV infusion of standard of care antibiotics and metronidazole for a total of 10 days. Dose based on postnatal age (PNA) and gestational age(GA)
  Arms: Group 4 (metronidazole)
Drug: metronidazole, clindamycin, or piperacillin-tazobactam — IV infusion of metronidazole, clindamycin, or piperacillin-tazobactam with scheduled CSF procedures per standard of care. Study drug will be given for for a total of 10 days. Dose based on postnatal age (PNA) and gestational age(GA)
  Arms: Group 5 (metronidazole/clindamycin/piperacillin-tazobactam)

SUMMARY:
The main purpose of this study is evaluate whether it is safe or not to use various combination of antibiotics (ampicillin, metronidazole, clindamycin, piperacillin-tazobactam, gentamicin) in treating infants with complicated intra-abdominal infections

DETAILED DESCRIPTION:
The most commonly used antibiotics in infants with complicated intra-abdominal infections are not labeled for use in this population because safety and efficacy data are lacking. This study will provide the safety information required for labeling. In addition, the pharmacokinetics(PK) and effectiveness data will also be collected during this study.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained from parent(s) or legal guardian(s) (Groups 1-5)
2. ≤33 weeks gestation at birth (Groups 1-3, 5)
3. ≥34 weeks gestation at birth (Groups 4 and 5)
4. PNA <121 days (Groups 1-5)
5. Sufficient venous access to permit administration of study drug (intravenous [IV]) (Groups 1-5)
6. Presenting physical, radiological, and/or bacteriological findings of a complicated intra-abdominal infection within 48 hours prior to randomization/first study drug dose (Groups 1-4)**. Complicated intra-abdominal infections include secondary peritonitis, NEC grade II or higher by Bell's criteria, Hirschsprung's disease with perforation, spontaneous intestinal perforation, meconium ileus with perforation, bowel obstruction with perforation, gastroschisis with necrosis and/or perforation, omphalocele with necrosis and/or perforation, neonatal appendicitis, intestinal pneumatosis or portal venous gas, free peritoneal air on abdominal radiographic examination, or abdominal abscess.
7. Suspected or confirmed infection for which the study drug may provide therapeutic benefit and planned CSF collection per standard of care (Group 5).

Exclusion Criteria*

1. History of anaphylaxis in response to study drugs (Groups 1-5)
2. Serum creatinine >2 mg/dL within 48 hours on measurement prior to and closest to randomization /first study drug dose (Groups 1- 5)**
3. Known ALT >250 U/L or AST >500 U/L on measurement closest to the time of randomization or first study drug dose (Groups 1-5)**
4. Any condition that, in the judgment of the investigator, precludes participation because it could affect participant safety (Groups 1-5)

   * Do not apply for Group 5 participants receiving drug per standard of care

     * Criteria must be satisfied by randomization (randomized Groups 1-3) or first study drug dose (non-randomized Groups 1-3, Group 4 and Group 5), whichever comes first.

Max Age: 120 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 260 (Actual)
Dates: Start 2013-12; Primary Completion 2017-01-15 (Actual); Study Completion 2017-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Micheal Cohen-Wolkowiez, MD, PhD, Principal Investigator — Duke University
Locations (50):
- United States (45):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arkansas Children's Hospital/Univ of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - Stanford University School of Medicine, Palo Alto, California
  - Rady Children's Hospital and Health Center, San Diego, California
  - University of California San Diego Medical Center, San Diego, California
  - Sharp Mary Birch, San Diego, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - University of Florida Jacksonville Healthcare, Inc., Jacksonville, Florida
  - Wolfson Children's Hospital, Shands Medical Center, Jacksonville, Florida
  - Georgia Regents University, Augusta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Riley Hospital, Indianapolis, Indiana
  - Wesley Medical Center, Wichita, Kansas
  - University of Kentucky Hospital, Lexington, Kentucky
  - Louisana State University Health Sciences Center, Shreveport, Louisiana
  - University of Maryland Hospital, Baltimore, Maryland
  - Floating Hospital for Children at Tufts Medical Center, Boston, Massachusetts
  - University of Minnesota Fairview University Medical Center, Minneapolis, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Kings County Hospital, Brooklyn, New York
  - Brookdale University Hospital, Brooklyn, New York
  - New York University School of Medicine, New York, New York
  - Columbia University Neonatology, New York, New York
  - Westchester Medical Center - New York Medical College, Valhalla, New York
  - University of North Carolina Hospital, Chapel Hill, North Carolina
  - Levine Children's Hospital, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - WakeMed Faculty Neonatology, Raleigh, North Carolina
  - New Hanover Reginal Medical Center, Wilmington, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Womens and Infant Hospital of Rhode Island, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Intermountain Medical Center, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
- Canada (5):
  - University of Alberta - Royal Alexandra Hospital, Edmonton, Alberta
  - University of British Columbia - British Columbia Women's Hospital, Vancouver, British Columbia
  - Manitoba Institute of Child Health, Winnipeg, Manitoba
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital Sainte-Justine, Montreal, Quebec

REFERENCES:
- [Derived] Smith MJ, Boutzoukas A, Autmizguine J, Hudak ML, Zinkhan E, Bloom BT, Heresi G, Lavery AP, Courtney SE, Sokol GM, Cotten CM, Bliss JM, Mendley S, Bendel C, Dammann CEL, Weitkamp JH, Saxonhouse MA, Mundakel GT, Debski J, Sharma G, Erinjeri J, Gao J, Benjamin DK Jr, Hornik CP, Smith PB, Cohen-Wolkowiez M; Best Pharmaceuticals for Children Act-Pediatric Trials Network Steering Committee. Antibiotic Safety and Effectiveness in Premature Infants With Complicated Intraabdominal Infections. Pediatr Infect Dis J. 2021 Jun 1;40(6):550-555. doi: 10.1097/INF.0000000000003034. PMID 33902072

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was enrolled but did not receive any dose of study drug. The participant is excluded from study result data analysis
Groups:
- Group 1: Ampicillin and gentamycin and metronidazole
  ampicillin and metronidazole and gentamicin: IV infusion of ampicillin and metronidazole and gentamicin for a total of 10 days. Dose based on postnatal age (PNA) and gestational age(GA)
- Group 2: ampicillin and gentamicin and clindamycin
  ampicillin and gentamicin and clindamycin: IV infusion of ampicillin and gentamicin and clindamycin for a total of 10 days. Dose based on postnatal age (PNA) and gestational age(GA)
- Group 3: piperacillin-tazobactam and gentamicin
  gentamicin and Piperacillin- tazobactam: IV infusion of gentamicin and Piperacillin- tazobactam for a total of 10 days. Dose based on postnatal age (PNA) and gestational age(GA)
- Group 4: Per standard of care antibiotics, and Metronidazole
  standard of care antibiotics and metronidazole: IV infusion of standard of care antibiotics and metronidazole for a total of 10 days. Dose based on postnatal age (PNA) and gestational age(GA)
- Group 5: metronidazole, clindamycin, or piperacillin-tazobactam
  metronidazole, clindamycin, or piperacillin-tazobactam: IV infusion of metronidazole, clindamycin, or piperacillin-tazobactam with scheduled CSF procedures per standard of care. Study drug will be given for for a total of 10 days. Dose based on postnatal age (PNA) and gestational age(GA)
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Started | 63 | 47 | 70 | 55 | 24
Completed | 28 | 12 | 23 | 9 | 22
Not Completed | 35 | 35 | 47 | 46 | 2

BASELINE CHARACTERISTICS:
Population: count of participants
  Note: the overall numbers above were based on "Per protocol population", defined as participants who received at least 1 study dose of each study drug of the enrolled treatment group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Total
Number analyzed (Participants) | 62 | 46 | 70 | 55 | 24 | 257
Age, Continuous [Mean (Standard Deviation); unit: Gestational Age (weeks)] | 27.3 (2.6) | 27.8 (3.0) | 27.5 (2.9) | 36.4 (2.1) | 28.9 (4.9) | 29.5 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 42 | 27 | 10 | 114
  Male | 44 | 29 | 28 | 28 | 14 | 143
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 11 | 11 | 12 | 1 | 47
  Not Hispanic or Latino | 46 | 34 | 52 | 38 | 20 | 190
  Unknown or Not Reported | 4 | 1 | 7 | 5 | 3 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1 | 0 | 2
  Asian | 0 | 1 | 1 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 20 | 10 | 23 | 8 | 6 | 67
  White | 32 | 26 | 37 | 35 | 14 | 144
  More than one race | 2 | 1 | 4 | 1 | 2 | 10
  Unknown or Not Reported | 7 | 8 | 5 | 9 | 2 | 31
Region of Enrollment [Number; unit: count of participants]
  Canada | 4 | 0 | 0 | 0 | 1 | 5
  United States | 58 | 46 | 70 | 55 | 23 | 252

OUTCOME MEASURES:

1. Primary Outcome: Death
Description: Number of Participants who experienced Death
Time Frame: Within 30 days after last dose of study drug, up to 40 days
Population: Full intent-to-treat population (patients who received at least 1 dose of any study drug)
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 63 | 47 | 70 | 56 | 24
Participants | 5 | 5 | 7 | 1 | 0

2. Secondary Outcome: Number of Participants With Therapeutic Success at Day 30
Description: Confirmed by 1).Alive, 2).Negative bacterial blood cultures, and 3). Clinical cure score >4.
  Clinical cure score =1 for each of the following elements:
  FiO2 ≤ baseline FiO2; Urine output ≥1 mL/kg/h for 24-hour period prior to assessment; Absence of inotropic support at time of assessment; Absence of mechanical ventilation at time of assessment; No seizure in 24-hour period prior to assessment; pH ≥7.25 or not measured in 24 hours prior to assessment
Time Frame: 30 days after last dose of study drug
Population: Participants who received at least 1 dose of each study drug. Does not apply to Group 5.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 62 | 46 | 70 | 55
Participants | 45 | 39 | 52 | 52

3. Other Pre Specified Outcome: Number of Participants With Feeding Intolerance
Description: Feeding intolerance confirmed by documentation of any feedings held for >24 consecutive hours in infants being fed
Time Frame: 90 days after last dose of study drug
Population: Participant who received at least 1 dose of each study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 62 | 46 | 70 | 55
Participants | 24 | 19 | 21 | 18

4. Other Pre Specified Outcome: Number of Participants With Grade 3 and/or Grade 4 Intraventricular Hemorrhage (IVH)
Description: Grade 3 IVH: Subependymal hemorrhage with extension into lateral ventricles with ventricular enlargement
  Grade 4 IVH: Intraparenchymal hemorrhage
Time Frame: 90 days after last dose of study drug
Population: Participant who received at least 1 dose of each study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 62 | 46 | 70 | 55
Participants | 2 | 4 | 4 | 0

5. Other Pre Specified Outcome: Number of Participants With Short Bowel Syndrome
Description: Short bowel syndrome: Operative reports documenting resection of bowel, estimated bowel length, and absence/presence of the ileocecal valve.
  Total parenteral nutrition for >42 consecutive days after bowel resection, or a residual small bowel length of less than 25% expected for gestational age
Time Frame: 90 days after last dose of study drug
Population: Participant who received at least 1 dose of each study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 62 | 46 | 70 | 55
Participants | 5 | 3 | 1 | 1

6. Other Pre Specified Outcome: Number of Participants With Intestinal Perforation
Description: Intestinal perforation: Radiological reports leading to the diagnosis of intestinal perforation. These include plain chest x-rays, plain abdominal x-rays, ultra-sonograms of the abdomen, contrast studies, and computed tomography scans of the abdomen and pelvis.
  Operative reports documenting surgical procedures leading to the diagnosis and/or treatment of intestinal perforation. These include placement of a surgical drain, laparotomy, intestinal resection, and ostomy placement
Time Frame: 90 days after last dose of study drug
Population: Participant who received at least 1 dose of each study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 62 | 46 | 70 | 55
Participants | 2 | 4 | 2 | 1

7. Other Pre Specified Outcome: Number of Participants With Intestinal Stricture
Description: Intestinal stricture: Radiology reports leading to the diagnosis of intestinal stricture. These include plain abdominal x-rays, upper gastrointestinal series with small bowel follow-through, contrast enema studies, and computed tomography scans of the abdomen and pelvis.
  Operative reports documenting surgical procedures leading to the diagnosis and/or treatment of intestinal stricture. These procedures include endoscopy, laparotomy, stricture dilatation, intestinal resection, and ostomy placement
Time Frame: 90 days after last dose of study drug
Population: Participant who received at least 1 dose of each study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 62 | 46 | 70 | 55
Participants | 3 | 2 | 4 | 1

8. Other Pre Specified Outcome: Number of Participants Progressed to a Higher Stage of Necrotizing Enterocolitis (NEC), if NEC is the Cause of the Complicated Intra-abdominal Infection
Description: Progression is determined by the clinical NEC scoring
Time Frame: 90 days after last dose of study drug
Population: Participant who received at least 1 dose of each study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 62 | 46 | 70 | 55
Participants | 1 | 2 | 0 | 1

9. Other Pre Specified Outcome: Number of Participants With Gastrointestinal Surgeries
Description: Determined by medical history and confirmed with hospital records. (Laparotomy)
Time Frame: 90 days after last dose of study drug
Population: Participant who received at least 1 dose of each study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 62 | 46 | 70 | 55
Participants | 27 | 15 | 26 | 10

10. Other Pre Specified Outcome: Number of Participants With Seizure
Description: documented seizure(s) in hospital records
Time Frame: 90 days after last dose of study drug
Population: Participant who received at least 1 dose of each study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 62 | 46 | 70 | 55
Participants | 4 | 0 | 2 | 1

11. Other Pre Specified Outcome: Number of Participants With Positive Blood Cultures
Description: Positive blood culture (bacterial or fungal)
Time Frame: 90 days after last dose of study drug
Population: Participant who received at least 1 dose of each study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 62 | 46 | 70 | 55
Participants | 8 | 4 | 12 | 5

ADVERSE EVENTS:
Time Frame: 90 days post last study dose
Description: Note: Participants who received at least 1 dose of any study drug in the randomized or assigned protocol treatment group were included in the intention-to-treat (ITT) population used for the safety and efficacy analyses
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
All-Cause Mortality (participants affected / at risk) | 5/62 | 5/46 | 7/70 | 1/55 | 0/24
Serious Adverse Events (participants affected / at risk) | 19/62 | 10/46 | 12/70 | 3/55 | 3/24
Other Adverse Events (participants affected / at risk) | 10/62 | 6/46 | 10/70 | 4/55 | 9/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=62) | Group 2 (N=46) | Group 3 (N=70) | Group 4 (N=55) | Group 5 (N=24)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinopathy of prematurity (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Necrotising colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Candida sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infantile apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Debridement (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Patent ductus arteriosus repair (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Extremity necrosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous occlusion (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=62) | Group 2 (N=46) | Group 3 (N=70) | Group 4 (N=55) | Group 5 (N=24)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (5) | 3 (3) | 4 (4) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 3 (7) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Intraventricular haemorrhage neonatal (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No